CLINICAL TRIAL: NCT01401296
Title: Evaluation of the Effectiveness of a Web-based Treatment Program for Depression (Deprexis) for the Reduction of Depressive Symptoms. A Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness of a Web-based Treatment Program for Depression for the Reduction of Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Deprexis
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: Depression; Online-Therapy; Deprexis; Self-help
MeSH Terms: conditions — Depression | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-list group (Active Comparator): Subjects receive access to deprexis after eight weeks
  Interventions: Behavioral: Wait-list
- Deprexis (Experimental): Web-based intervention deprexis consists of ten online modules (plus one introductory and one summary module) representing different psychotherapeutic strategies with a strong focus on evidence-based cognitive-behavioral techniques (e.g. interpersonal skills). Each module lasts approximately 10-60 minutes (e.g. depending on the user´s reading speed). Modules are sequential and organized as simulated dialogues. Each module refers and builds upon previous one. The program is delivered at no cost to participants.
  Interventions: Behavioral: Deprexis

INTERVENTIONS:
Behavioral: Deprexis — Behavioral: Deprexis (10 sessions) delivered online versus wait-list control group
  Other Names: web-based treatment program for depression
  Arms: Deprexis
Behavioral: Wait-list — Behavioral: the wait-list group receives Deprexis after 8 weeks
  Other Names: web-based treatment for depression after 8 weeks
  Arms: Wait-list group

SUMMARY:
200 persons with depression are recruited via internet depression forums devoted to depression and are randomly assigned either to the online program deprexis or to a wait-list control condition. All participants receive free-of-charge online access to deprexis either immediately or with an eight week delay.

Prior to intervention and eight weeks later, both groups are assessed via an anonymous online survey which was implemented using the software package OPST®. The survey consists of different questionnaires. The Beck Depression Inventory (BDI) represents the primary outcome. It is assumed that the severity of depressive symptoms will improve to a significantly greater extent in the deprexis than in the wait-list control condition in the course of eight weeks.

DETAILED DESCRIPTION:
Deprexis is a web-based intervention that can be obtained online (www.deprexis.com). Deprexis encompasses 10 content modules with a strong focus on evidence-based cognitive-behavioral techniques, either from its so-called first (behavior-oriented), second (cognitive-oriented) or third wave (e.g. mindfulness and acceptance): (1) psychoeducation, (2) behavioral activation, (3) cognitive modification, (4) mindfulness and acceptance, (5) interpersonal skills, (6) relaxation, physical exercise and lifestyle modification, (7) problem solving and (8) expressive writing and forgiveness, (9) positive psychology and (10) dreamwork and emotion-focus interventions. The ten modules are framed by one introductory and one summary module. Communication is carried out online via simulated dialogues. Patients have to respond to narrative text messages from the virtual therapists in multiple-choice response fashion, enabling them to express doubt, to affirm a particular message or to request more information. Text messages are aided with drawings, photographs and animations. The program is adaptive and selects exercises and contents on the basis of the subject's response. The modules are sequential and each module refers and builds upon previous one. Modules can (and should be) repeated within the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* registration in a moderated online forum exclusively for affective disorders
* (externally) confirmed diagnosis of a unipolar depression
* informed consent (provided online in line with regulations by the Hamburg Department of Data Security)

Exclusion Criteria:

* unable to provide informed consent
* diagnosis of bipolar or schizophrenia spectrum disorders
* substantial neurological impairment (e.g. dementia)
* acute suicidal tendencies as assessed with the Suicide Behaviors Questionnaire-Revised (SBQ-R). Subjects excluded for this reason are provided various emergency contacts and phone numbers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Severity of depressive symptoms | 7 Days
  Severity of depressive symptoms as assessed with the Beck Depression Inventory (BDI)

SECONDARY OUTCOMES:
quality of life as assessed by the WHO Quality of Life scale (WHO-QOL BREF) | 7 days
  The WHO-QOL- Bref is an abbreviated 26-item version of the WHO-QOL-100 which covers four domains of quality of life (QoL): physical. psychological. social. environment.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Mortz, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- See also: link to metacognitive training site, where training material can be downloaded cost-free — http://www.deprexis.com